CLINICAL TRIAL: NCT06568874
Title: Effect of Virtual Reality Versus Conservative Treatment in Sensorimotor Function of Upper Extremity in Chronic Stroke Patients
Brief Title: Effect of VR Versus CT in Sensorimotor Function of Upper Extremity in Chronic Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/740
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exp Group (Experimental)
  Interventions: Combination Product: Virtual Reality (VR) Therapy
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Conservative Treatment

INTERVENTIONS:
Combination Product: Virtual Reality (VR) Therapy — Intervention: Patients in this group will receive therapy using VR technology. This involves engaging in various sensorimotor training exercises and tasks in an immersive virtual environment. The VR sessions are designed to be interactive and adaptive, providing real-time feedback to the user. The exercises will target the improvement of motor functions, coordination, and strength of the affected upper extremity.
  Duration and Frequency: The specific regimen may involve sessions several times a week, with each session lasting between 30 to 60 minutes, over a period of several weeks or months, depending on the study design.
  Arms: Exp Group
Diagnostic Test: Conservative Treatment — Intervention: Patients in this group will receive traditional rehabilitation therapies, which may include:
  Physical Therapy (PT): Exercises and activities aimed at improving strength, flexibility, and coordination of the upper limb.
  Occupational Therapy (OT): Functional task training to enhance daily living skills and independence, focusing on the use of the upper extremity.
  Manual Therapy: Techniques such as massage or joint manipulation to improve mobility and reduce pain.
  Home Exercise Programs: Prescribed exercises to be performed at home to reinforce therapy sessions.
  Duration and Frequency: Similar to the VR group, this regimen may involve regular sessions several times a week, with each session lasting between 30 to 60 minutes, over a comparable period.
  Arms: Control Group

SUMMARY:
Virtual reality (VR) therapy has shown promising results in improving sensorimotor function of the upper extremity in chronic stroke patients compared to conservative treatments. VR offers immersive, interactive environments that can enhance motivation and engagement in rehabilitation exercises.

ELIGIBILITY:
Inclusion Criteria

* Patients with a confirmed diagnosis of chronic stroke (at least 6 months post-stroke).

Age:

* Upper Extremity Impairment:
* Ability to provide informed consent to participate in the study.

Exclusion Criteria

* Severe communication difficulties that would impede the ability to follow instructions during therapy.
* Severe spasticity in the affected upper limb (Modified Ashworth Scale score of 4 or higher).
* Other Neurological Conditions

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) for Upper Extremity | 12 Months
  The Fugl-Meyer Assessment (FMA) for Upper Extremity is a widely used and validated tool to evaluate motor function, balance, sensation, and joint functioning in individuals who have had a stroke. It specifically assesses the sensorimotor function of the upper extremities.
  Scoring:
  The upper extremity section of the FMA includes 33 items, each scored on a scale of 0 to 2:
  0: Cannot perform
  1. Performs partially
  2. Performs fully The maximum score for the upper extremity section is 66, indicating optimal function.
Stroke Impact Scale (SIS) | 12 months
  The Stroke Impact Scale (SIS) is a self-report questionnaire that evaluates the impact of stroke on multiple dimensions, including strength, hand function, activities of daily living (ADL), mobility, communication, emotion, memory, thinking, and participation.
  Each item is scored on a scale of 1 to 5:
  1: Unable to do 5: Not difficult at all Higher scores indicate a lesser impact of stroke on the patient's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital,Shadman 1, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No